CLINICAL TRIAL: NCT06506734
Title: Prevalence of Dental Dyschromia and Impact on the Quality of Life of Participants with Prolonged Hyperbilirubinemia During Their Early Years
Brief Title: Dental Dyschromia and Quality of Life in Early Prolonged Hyperbilirubinemia
Acronym: SMILE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0443
Record Dates: First submitted 2024-06-28; First posted 2024-07-17 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Dental Diseases
Keywords: Hyperbilirubinemia; Biliary Atresia; Progressive Familial Intrahepatic Cholestasis (PFIC); Alagille Syndrome; Tooth Discoloration
MeSH Terms: conditions — Stomatognathic Diseases; Hyperbilirubinemia; Biliary Atresia; Cholestasis, progressive familial intrahepatic 1; Alagille Syndrome; Tooth Discoloration | interventions — Surveys and Questionnaires; Moire Topography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dental Dyschromia in Hyperbilirubinemia Patients: 30 minutes
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — * " Psychosocial Impact of Dental Aesthetics Questionnaire " PMID 24280547
  * " Orofacial Esthetic Scale " PMID 30856637
  * " Orofacial Esthetic Scale " PMID 34231057
  * A photograph of the patient's smile will be sent to 2 dentists who will also assess the presence or absence of dental dyschromia.
  Other Names: Photograph

SUMMARY:
The main objective of this study is to assess the prevalence of dental discoloration (dental dyschromia) in children who experienced high levels of bilirubin in their blood (hyperbilirubinemia) during their early years. The study will also examine risk factors associated with this condition, such as the duration and severity of hyperbilirubinemia, underlying diseases, and treatments received.

The researchers hypothesize that the quality of life of individuals with dental dyschromia is lower than that of individuals without dyschromia. The results of this study will be used to discuss coverage for dental care with health insurance for children affected by this condition.

ELIGIBILITY:
Inclusion Criteria:

* A patient with biliary atresia, progressive familial intrahepatic cholestasis, or Alagille syndrome
* Patient or legal representative not opposed to participating in this research.

Exclusion Criteria:

* Inability to understand and respond to quality of life questionnaires

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 12 to 18 years
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-02 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dental dyschromia | from birth to study completion, a maximum of 19 years
  presence of dyschromia or not evaluated by 2 investigators

SECONDARY OUTCOMES:
Presence or absence of dental dyschromia | through study completion, an average of 18 months
  Presence or absence of dental dyschromia based on various variables such as bilirubin levels or the duration of hyperbilirubinemia.

OTHER OUTCOMES:
Quality of life score by patient group | through study completion, an average of 18 months
  Assess the quality of life score based on the patient's group classification

CONTACTS AND LOCATIONS:
Overall Officials: Nolwen LABORDE, MD, Principal Investigator — University Hospital, Toulouse
Locations (9):
- France (9):
  - University Hospital Bordeaux, Bordeaux
  - University Hosptial Caen, Caen
  - University Hospital Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - University Hospital Marseille, Marseille
  - Assistance Publique-Hôpitaux de Paris, Hôpital Bicêtre, FHU Hépatinov, Paris
  - Assistance Publique-Hôpitaux de Paris, Hôpital Bretonneau, Paris, Paris
  - Assistance Publique-Hôpitaux de Paris, Hôpital Necker, Paris
  - University Hospital Rennes, Rennes